CLINICAL TRIAL: NCT04299529
Title: Urinary Proteomics Combined With Home Blood Pressure Telemonitoring for Health Care Reform: a Randomised Controlled Trial
Brief Title: Urinary Proteomics Combined With Home Blood Pressure Telemonitoring for Health Care Reform
Acronym: UPRIGHT-HTM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Collaborators: Alliance for the Promotion of Preventive Medicine (Unknown)
Responsible Party: Principal Investigator, Jan A. Staessen, Professor of Medicine, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: UPRIGHT-HTM, version 4.0
Record Dates: First submitted 2020-03-02; First posted 2020-03-06 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Protein Deregulation; Blood Pressure; Health Care Utilization; Cost Effectiveness; Patient Empowerment
MeSH Terms: conditions — Patient Acceptance of Health Care; Patient Participation

STUDY DESIGN:
Intervention Model Description: Parallel group design
Who Masked: Outcomes Assessor
Masking Description: Caregivers will know the group to which their patients were randomly assigned. In the two groups, both patients and caregivers will have full access to the HTM data. In both treatment groups, caregivers will be informed about the UPP risk profile. However, in the experimental group, patients will be informed about their UPP risk profile shortly after randomisation and in the control group, only when they leave randomised follow-up or at the completion of the trial. The central study coordinating team will remain blinded to the primary endpoint and all of its components until completion of the trial and until all datasets have been cleaned and frozen for the final analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HTM plus UPP (Experimental): Urinary proteomic profiling administered on top of home blood pressure telemonitoring and guideline-endorsed non-pharmacological and pharmacological management of risk factors
  Interventions: Diagnostic Test: In-vitro urinary diagnostic test
- HTM alone (Other): Home blood pressure telemonitoring administered on top of non-pharmacological and pharmacological management of risk factors
  Interventions: Diagnostic Test: In-vitro urinary diagnostic test

INTERVENTIONS:
Diagnostic Test: In-vitro urinary diagnostic test — Urinary proteomic profiling (UPP) using established multidimensional urinary markers for progression to CKD (CKD273), left ventricular dysfunction (HF1 and HF2) and coronary heart disease (CAD238 and ACSP75) - in-vitro test certified in Germany and by extension in the EU (DE/CA09/0829/IVD/001, DE/CA09/0829/IVD/005).

SUMMARY:
UPRIGHT-HTM will compare risk stratification, treatment efficiency and health economic outcomes of a diagnostic approach based on home blood pressure telemonitoring combined with urinary proteomic profiling with home blood pressure telemonitoring alone

DETAILED DESCRIPTION:
Hypertension is by far the dominant reversible risk factor dwarfing most others in the pathogenesis of chronic kidney disease (CKD) and diastolic left ventricular dysfunction (DVD), two archetypes of chronic age-related diseases, which are rampant in ageing societies in epidemiological transition. Home blood pressure telemonitoring (HTM) is a recommended approach in the diagnosis and management of hypertension. Urinary peptidomic profiling (UPP) holds great promise in individualising prevention and treatment of CKD and DVD and associated complications, such as coronary heart disease. Making use of these modern technologies, UPRIGHT-HTM is an investigator-initiated randomised clinical trial with a patient-centred design, for the first time, comparing HTM combined UPP (experimental group) to HTM alone (control group) in risk profiling and as guide to starting or intensifying management of risk factors to prevent established disease. The trial will run in Europe, sub-Saharan Africa and South America. Eligible patients, aged 55-75 years old, are asymptomatic, but have three or more CKD- or DVD-related risk factors, preferably including hypertension, type 2 diabetes mellitus, or both, and do have internet skills. The primary endpoint consists of a composite of new-onset intermediate endpoints (microalbuminuria, progression of CKD, diabetic or hypertensive retinopathy, electrocardiographic or echocardiographic left ventricular hypertrophy or DVD and hard outcomes (cardiovascular mortality and non-fatal complications, including myocardial infarction, heart failure and stroke). Secondary objectives are demonstrating that combining HTM with UPP is feasible and cost-effective in a multicultural context, defining the molecular signatures of early CKD and DVD, and with help of stakeholders educating and empowering patients. Assuming an accrual time of 1 year, a median follow-up of 4 years, a 10% dropout rate, a 20% risk of the primary endpoint in the control group and 30% risk reduction in the experimental group, requires 1000 patients to be randomised in a 1:1 proportion with the two-sided alpha level and power set 0.05 and 0.80, respectively. The expected outcome is proving the superiority in terms of efficiency and cost-effectiveness of HTM combined with UPP vs HTM alone, which should lead to redesigning the clinical workflow, putting greater emphasis on preventing rather than curing established disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have at least three additional guideline-defined risk factors, preferably including hypertension, type 2 diabetes mellitus (T2DM), or both;
* Patients should be willing patients to engage for the duration of the study in home blood pressure telemonitoring (1 reading per day);
* Patients must have an email address and internet access via smartphone, tablet, or laptop or desktop computer;
* Patients should comply with the study protocol during the run-in phase.

Exclusion Criteria:

* Type 1 diabetes mellitus;
* Absence of a practicable echocardiographic window;
* Previous or concurrent severe cardiovascular or non-cardiovascular disease;
* Cancer within 5 years of enrolment;
* Suspected substance abuse;
* Psychiatric illness;
* Use of nephrotoxic drugs;
* Particpation in another clinical study.

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2020-04-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Primary composite endpoint | After a run-in period of 2 to 5 weeks to check the eligibility, patients will be randomized and followed up for 4 years
  The primary endpoint is a composite of intermediary and "hard" cardiovascular-renal endpoints.
  The "intermediate endpoints" are diabetic nephropathy, progression to a higher CKD stage, doubling of serum creatinine, an eGFR decrease by 30% or more or eGFR declining below 45 ml/min/1.73 m2, new-onset hypertensive or diabetic retinopathy, electrocardiographic or echocardiographic left ventricle hypertrophy, and diastolic left ventricular dysfunction.
  The "hard" composite cardiovascular endpoint includes cardiovascular mortality, and nonfatal myocardial infarction, nonfatal hospitalised heart failure, and nonfatal stroke, not including transient ischemic attack. The "hard" renal outcomes include macroalbuminuria, the need for renal-replacement therapy, and death to renal causes.
Change in serum creatinine (mg/dl) | After a run-in period of 2 to 5 weeks to check the eligibility, patients will be randomized and followed up for 4 years
  The concentration of creatinine in serum, expressed in mg/dl, will be measured, using Jaffe's method with modifications () in certified laboratories applying isotope-dilution mass spectrometry for calibration (Clin Chem 2006; 52: 5-18).
Change in eGFR (ml/min/1.73m2) | After a run-in period of 2 to 5 weeks to check the eligibility, patients will be randomized and followed up for 4 years
  eGFR will be derived from the serum creatinine concentration by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation (Ann Intern Med 2009; 150: 604-612) and expressed in ml/min/1.73 m2.
Progression of CKD | After a run-in period of 2 to 5 weeks to check the eligibility, patients will be randomized and followed up for 4 years
  The National Kidney Foundation Kidney Disease Outcomes Quality Initiative guideline will be followed (Kidney Int Suppl 2013;3:1-150): eGFR ≥90, 60-89, 45-59, 30-44, 15-29 and <15 mL/min/1.73 m2 for Stage 1, 2, 3A, 3B, 4 and 5, respectively
Incidence of diabetic nephropathy | After a run-in period of 2 to 5 weeks to check the eligibility, patients will be randomized and followed up for 4 years
  Microalbuminuria of 30 microgram per gram creatinine or more in two of three morning urine samples collected on three consecutive days.
Incidence of diabetic retinopathy | After a run-in period of 2 to 5 weeks to check the eligibility, patients will be randomized and followed up for 4 years
  Non-proliferative diabetic retinopathy (NPDR): early NPDR, at least one microaneurysm ; moderate NDPR, characterized by multiple microaneurysms, dot-and-blot hemorrhages, venous beading, and/or cotton wool spots; severe NPDR, diffuse intraretinal hemorrhages and microaneurysms in four quadrants, venous beading in two or more quadrants, or severe intraretinal microvascular abnormalities
  Proliferative diabetic retinopathy (PDR): fibrovascular proliferation extending beyond the internal limiting membrane; vitreous hemorrhage; retinal detachment, macular edema
  (https:// https://webeye.ophth.uiowa.edu/eyeforum/tutorials/Diabetic-Retinopathy-Med-Students/Classification.htm)
Incidence of hypertensive retinopathy | After a run-in period of 2 to 5 weeks to check the eligibility, patients will be randomized and followed up for 4 years
  Grade 1: mild narrowing and tortuosity of the retinal arterioles; Grade 2: definite focal retinal arteriolar narrowing and arteriovenous nipping; Grade 3: retinal hemorrhages and cotton wool spots; Grade 4: papilledema
Incidence of electrocardiographic LV hypertrophy | After a run-in period of 2 to 5 weeks to check the eligibility, patients will be randomized and followed up for 4 years
  The Sokolow-Lyon index is the sum of the S-wave in V1 and the R wave in V5 or V6, whichever is greater; the threshold value is 3.5 mV (PMID 31352838, 19015402, 28789616); in regularly calibrated ECGs, 1 mV is 10 mm along the vertical axis;
  The Cornell product is the sum of RaVL and RV5 with 6 mV added for women, multiplied by the QRS duration in milliseconds; the cut-off value is 2440 mV × ms (PMID 31352838, 19015402, 28789616);
  Increased R-wave in aVL: the threshold values is 1.1 mV;
  ST segment down sloping in V4-V6 with T-top inversion.
  Based on these criteria the investigators will classify patients as having or not having electrocariographic LV hypertrophy
Incidence of echocardiographic LV hypertrophy | After a run-in period of 2 to 5 weeks to check the eligibility, patients will be randomized and followed up for 4 years
  Guidelines should be applied for acquisition and off-line analysis of the echocardiographic imaging studies (PMID 15452478, 19187853, 27037982); LV mass will be calculated using a formula validated by necropsy (PMID 2936235, 15452478); LVM = 0.8 × (1.04 × (EDD + IVS + LPW)3 - EDD)3) + 0.6; expressed in gram; LV mass will be indexed to body surface; the threshold values are ≥95/≥115 g/m2 in women/men.
Incidence of diastolic LV dysfunction | After a run-in period of 2 to 5 weeks to check the eligibility, patients will be randomized and followed up for 4 years
  Diastolic LV dysfunction will be defined as an abnormally low age-specific transmitral E/A ratio, indicative of impaired relaxation, or a mildly-to-moderately elevated left ventricular filling pressure (E/e' >8.5) with normal or decreased age-specific E/A ratio. The ejection fraction should be over 50% (Circ Heart Fail 2009;2: 105-112).
Incidence of CV mortality | After a run-in period of 2 to 5 weeks to check the eligibility, patients will be randomized and followed up for 4 years
  ICD10 codes I00-I99
Incidence of nonfatal myocardial infarction | After a run-in period of 2 to 5 weeks to check the eligibility, patients will be randomized and followed up for 4 years
  ICD10 codes I21,I22
Incidence of nonfatal heart failure | After a run-in period of 2 to 5 weeks to check the eligibility, patients will be randomized and followed up for 4 years
  ICD10 code I50
Incidence of nonfatal stroke | After a run-in period of 2 to 5 weeks to check the eligibility, patients will be randomized and followed up for 4 years
  ICD10 codes I60-I63
Incidence of CKD | After a run-in period of 2 to 5 weeks to check the eligibility, patients will be randomized and followed up for 4 years
  ICD10 codes N17, N18

SECONDARY OUTCOMES:
EQ-5D (scale ranging from 0 [worst possible] to 100 [best possible]) | After a run-in period of 2 to 5 weeks to check the eligibility, patients will be randomized and followed up for 4 years.
  Quality of life will be assessed using the EQ-5D quality of life questionnaire (http://www.euroqol.org)
Health-economic analysis | After a run-in period of 2 to 5 weeks to check the eligibility, patients will be randomized and followed up for 4 years.
  For health-economic evaluation, the EQ-5D patient-administered questionnaire (https://www.euroqol.org) is of particular importance, as Quality Adjusted Life Years (QALYs) can be generated from this simple instrument

CONTACTS AND LOCATIONS:
Overall Officials: Lutgarde Thijs, MSc, Principal Investigator — University of Leuven
Locations (12):
- Belgium (3):
  - European Kidney Health Aliance, Brussels
  - Diabetes Liga, Ghent
  - Alliance for the Promotion of Preventive Medicine, Mechelen
- Steno Diabetes Center Copenhagen, Gentofte Municipality, Denmark
- Mosaiques-Diagnoostics and Therapeutics AG, Hanover, Germany
- Biomedical Research Foundation of the Academy of Athens, Athens, Greece
- Department of Internal Medicine, Faculty of Clinical Sciences, College of Health Sciences, University of Abuja, Abuja, Nigeria
- Poland (2):
  - Department of Hypertension, Medical University of Gdańsk, Gdansk
  - First Department of Cardiology, Interventional Electrocardiology and Hypertension, Jagiellonian University Medical College, Krakow
- Department of Internal Medicine, Division of Hypertension, University Medical Centre Ljubljana, Ljubljana, Slovenia
- Hypertension in Africa Research Team, Medical Research Council Unit for Hypertension and Cardiovascular Disease, North-West University, Potchefstroom, South Africa
- Centro de Nefrología and Departamento de Fisiopatología, Hospital de Clínicas, Universidad de la República, Montevideo, Uruguay

IPD SHARING:
Plan to Share IPD: Yes
A motivated request for data transfer for scientific purposes should be addressed to Prof Jan A. Staessen
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Starting after completion of the trial for a duartion of 5 years
Access Criteria: Approval by the Ethics Committee of the University Hospitals Leuven

REFERENCES:
- [Derived] Chori BS, An DW, Martens DS, Yu YL, Gilis-Malinowska N, Abubakar SM, Ibrahim EA, Ajanya O, Abiodun OO, Anya T, Tobechukwu I, Isiguzo G, Cheng HM, Chen CH, Liao CT, Mokwatsi G, Stolarz-Skrzypek K, Wojciechowska W, Narkiewicz K, Rajzer M, Brguljan-Hitij J, Nawrot TS, Asayama K, Reyskens P, Mischak H, Odili AN, Staessen JA; UPRIGHT-HTM Investigators. Urinary proteomics combined with home blood pressure telemonitoring for health care reform trial-First progress report. J Clin Hypertens (Greenwich). 2023 Jun;25(6):521-533. doi: 10.1111/jch.14664. Epub 2023 May 6. PMID 37147930